CLINICAL TRIAL: NCT04740528
Title: Department of Nutrition Science, Medical Faculty, Universitas Diponegoro Semarang, Indonesia
Brief Title: Preference of Protein Intake and FTO rs1558902 Gene Polymorphism Among Women Obese
Status: Completed | Type: Observational
Sponsor: Universitas Diponegoro (Other)
Responsible Party: Principal Investigator, Etika Ratna Noer, Department of Nutrition, Medical Faculty, Universitas Diponegoro
Other Study IDs: FTO
Record Dates: First submitted 2021-02-01; First posted 2021-02-05 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2021-02

CONDITIONS: Obesity Adult Onset
Keywords: woman Obese; fto-gen; rs1558902; protein intake

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — whole blood specimen intravenous 5ml
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: fto gene testing — Blood samples were collected after a 12-h fasting by Prodia Laboratory for DNA isolation and biochemical analysis

SUMMARY:
The concept personalized gene-based nutrition combines genetic information with specific dietary intake that is crucial in managing obesity. Obesity experienced by adult women is generally caused by inapproriate diet and sedentary lifestyle. Variations in the fat mass and obesity-related gene (FTO) has been linked with susceptibility to obesity, but diet seems to change the relationship. A single nucleotide polymorphism (SNP) in the fat mass and obesity-associated gene (FTO) is a potent predictor of human obesity. Higher protein diets were more appropriate than standard protein diets, and frequently recommended as a weight loss plan as it prevents the loss of lean tissue mass. Nevertheless, high intakes of proteins may adversely affect metabolic functions. Multi studies have explored associated FTO polymorphisms with obesity in different populations. However, the contribution of the FTO common variants to obesity is controversial in Asian people, some studies showed rs1558902 was statistically associated with BMI, but other results reported FTO gene is not statistically associated with obesity. Given the diversity of Asian populations, the investigators generated a hypothesis whether relations between preference protein intake and FTO rs1558902 gene polymorphism exist in selected Indonesian obesity women

DETAILED DESCRIPTION:
The sample size was calculated based on the difference in the proportion of variation of the gene FTO rs1558902 allele A between obese participants, which previous study estimated to be approximately 6% for populations from Malaysia. Using a power of 80% and a level of significance of 5%, the investigators required 100 obese participants.

BMI and body fat which were assessed by SECA body analyzer (SECA 201). Blood samples were collected after a 12-h minimum fast by Prodia Laboratory for DNA isolation and biochemical analysis

ELIGIBILITY:
Inclusion Criteria:

* Body Mass index > 25 kg/m2
* waist circumference > 80 cm

Exclusion Criteria:

* chronic disease
* have pregnancy
* consume diet supplement, drugs

Ages: 35 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: healthy woman obese and pre menopause
Sampling Method: Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
fto gene rs 1558902 | day 1
  Genomic DNA was extracted from 300 ml of buffy coat using spin colomn method. rs 1558902 were genotyped using TaqMan probes C__30090620_10
interleukin-6 | day 1
  plasma IL-6 was determined by enzyme-linked immunosorbent method (EliKine™ Human IL-6 ELISA Kit)

CONTACTS AND LOCATIONS:
Overall Officials: Etika Noer, PhD, Principal Investigator — Diponegoro University
Locations (1):
- Etika Ratna Noer, Semarang, Central Java, Indonesia